CLINICAL TRIAL: NCT04077385
Title: A Novel, Memory-Updating Technique to Attenuate Responding to High Calorie Food Cues, Food Intake, and Body Weight Among Individuals With Overweight/Obesity
Brief Title: Memory-Updating Technique to Reduce Food Craving and High Calorie Food Intake Among Individuals With Overweight/Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI resigned from faculty position and K23 award was terminated early
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lisa J Germeroth, PhD, Assistant Professor, Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY18100137; 1K23DK117994-01 (NIH)
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Overweight; Obesity; Craving; Eating Behavior
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This study uses a two-arm parallel assignment in which participants are randomized to either a high calorie food retrieval + high calorie food extinction (R-E training) group or to a non-food retrieval + high calorie food extinction (extinction control) group.
Masking Description: There will not be masking in the current study for participants as they will know if they are observing either high calorie pictorial food cues or non-food-related pictorial cues during the retrieval portion of the R-E/extinction training days. The investigator will also not be masked given that participants will be observed completing the R-E training task during sessions to ensure compliance, which involves observing participants advance through the task via a mirrored image on a second desktop monitor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrieval Extinction (R-E) Training Group (Experimental): On the two retrieval-extinction (R-E)/extinction training days, participants randomized to the R-E training group will observe 5-min of high calorie pictorial food cues during "retrieval" which will purportedly retrieve cue-reward associative memories. This will be followed by 60-min of extinction training to high calorie food cues. The R-E training group will only differ from the extinction control group in regards to the 5-min exposure to high calorie food cues prior to the 60-min of extinction training to high calorie food cues.
  Interventions: Behavioral: Retrieval-extinction (R-E) Training
- Extinction Control Group (Active Comparator): On the two retrieval-extinction (R-E)/extinction training days, participants randomized to the extinction control group will observe 5-min of non-food-related cues (e.g., pictures of office supplies, tools) during "retrieval," which will purportedly avoid retrieval of the food cue-reward associative memories that are targeted in the R-E training group. The 5-min of exposure to non-food-related cues will be followed by the same 60-min of extinction training to high calorie food cues that the R-E training group receives.
  Interventions: Behavioral: Extinction Training

INTERVENTIONS:
Behavioral: Retrieval-extinction (R-E) Training — The retrieval-extinction (R-E) training intervention will occur on two consecutive days and consist of (a) retrieval of high calorie food cue-reward associative memories and (b) 60-min extinction training for high calorie foods. During the 5-min of retrieval, participants will observe 30 high calorie food images (e.g., cakes, cookies, muffins, hamburgers, french fries, potato chips, pizza). Images will be presented in E-Prime for 8-s each (2-s delay between images). After the 5-min of retrieval and a 10-min rest period, participants will engage in 60-min of extinction training for high calorie foods consisting of 12, 5-min high calorie food cue sequences: 6 image sequences and 6 real food sequences. The real foods will consist of a small portion of high calorie snack foods such as a single M&M or potato chip.
  Arms: Retrieval Extinction (R-E) Training Group
Behavioral: Extinction Training — The extinction control group will engage in two consecutive days of intervention consisting of (a) retrieval of memories not associated with high calorie foods and (b) 60-min extinction training for high calorie foods. During the 5-min of retrieval, participants will observe 30 non-food-related neutral images (e.g., office supplies, tools). Images will be presented in E-Prime for 8-s each (2-s delay between images). After the 5-min of retrieval and a 10-min rest period, participants will engage in 60-min of extinction training for high calorie foods consisting of 12, 5-min high calorie food cue sequences: 6 image sequences and 6 real food sequences. The real foods will consist of a small portion of high calorie snack foods such as a single M&M or potato chip. The 60-min extinction training is the same as the extinction training received by participants in the R-E training intervention.
  Arms: Extinction Control Group

SUMMARY:
This study will evaluate the effects of retrieval-extinction (R-E) training on responding to high calorie foods including self-report craving, physiological responding, and high calorie food intake in adults with overweight/obesity. R-E training aims to update the memories that associate cues (i.e., high calorie food) with reward (i.e., consumption). R-E training involves "retrieving" these cue-reward associative memories through brief presentation of relevant cues, resulting in instability of the memories and providing an opportunity to be updated via reconsolidation. Presenting relevant cues while not allowing consumption (i.e., extinction training) during reconsolidation can modify the unstable cue-reward memories, resulting in lasting reductions of craving and intake. This study will be the first to test the effects of R-E training on craving for and intake of high calorie foods in humans. To examine the effects of R-E training on food craving, physiological response (heart rate, skin conductance, salivation), and food intake, 150 adults with overweight/obesity will complete baseline food cue-reactivity and intake tasks in the lab. Participants will be randomized to observe high calorie food cues (i.e., "retrieval" of food cue-reward memories; R-E training group) or non-food cues (i.e., no retrieval of food cue-reward memories; extinction control group) and engage in 60 min of extinction training for high calorie foods. R-E/extinction control training will occur on two consecutive days and four follow-up food cue-reactivity sessions through 3 months. Weight will be assessed at each session and in-lab food intake at 1- and 3-months. Recent food/drink intake will also be assessed at each session. Some participants (n=75) will complete a pilot portion of the study involving real-world data collection of naturally-occurring food cues, craving, and food intake via smartphone. It is hypothesized that: (1) R-E training (vs. extinction control) will decrease high calorie food cue-reactivity (self-report craving, heart rate, skin conductance, salivation) and intake assessed in the lab, as well as self-report craving and food intake assessed in the real world; and (2) decreased high calorie food cue-reactivity will be a mechanism through which R-E training reduces high calorie food intake at follow-up. The Principal Investigator will explore associations between lab and real-world cue-elicited craving and food intake, and the effect of R-E training on weight.

DETAILED DESCRIPTION:
Participants (N=150) with overweight/obesity (body mass index ≥25.0 kg/m^2) will be recruited locally via media outlets, flier postings, and local research registries to participate in a novel laboratory-based intervention to attenuate craving for and intake of high calorie foods. Interested individuals will be screened over the phone to determine eligibility to participate. Once participants are deemed eligible, they will be scheduled for their sessions. All participants will attend seven sessions, the first four of which occur on four consecutive days: a baseline cue-reactivity session, two consecutive days of either retrieval extinction (R-E) training or extinction control, and four follow-up food cue-reactivity sessions taking place 24-hr, 2-weeks, 1-month, and 3-months after the second R-E/extinction training control session. Participants in the latter half of study recruitment will also participate in ecological momentary assessment (EMA) to collect data on real-world food cues, craving, and food intake. Those participants will engage in one pre-baseline session to receive instructions and a tutorial on a run-in period of baseline EMA data collection prior to the baseline session. Participants will be food-deprived for three hr prior to all sessions to standardize hunger. Participants will also be asked to avoid consuming high calorie foods/drinks from the night before the baseline session through the end of the day of the 24-hr follow-up session to avoid reinforcing high calorie food intake before or after extinction.

BASELINE SESSION: At the 2.5-hr baseline session, participants will first provide written Institutional Review Board (IRB)-approved informed consent. Participants will then be interviewed to report recent food/drink intake as well as various health-related behaviors (nicotine, alcohol, caffeine, cannabis, and other substance use, medication use, sleep, physical activity). Next, after a 10-min acclimation period, participants will complete baseline assessments of hunger and craving, including self-report state food craving, skin conductance, heart rate, and salivation. To assess heart rate, electrodes will be placed beneath the ribcage and the clavicle.Two silver/silver chloride (Ag/AgCl) electrodes will be affixed to the palm of the non-dominant hand to assess skin conductance. Heart rate and skin conductance will be assessed and scored using MindWare Technologies hardware and MindWare Technologies/BioLab software. The Strongin-Hinsie Peck procedure will be used to assess saliva production. Three pre-weighed cotton dental rolls, one placed beneath the tongue and two placed buccally for two min, will be removed and placed in plastic bags for weighing to assess the amount of saliva secreted. Participants will then complete a food cue-reactivity task using E-Prime software and a bogus taste test (see "TASK DESCRIPTION" section below). At the end of the session, participants will complete measures of demographics (e.g., age, sex, race), socioeconomic status, motivation to lose weight, trait food craving, dietary restraint and disinhibited eating, impulsivity, negative and positive affect, depressive symptoms, social support, food insecurity, sleep, physical activity, disordered eating symptoms, eating behaviors, reward-based eating drive, weight and diet history, and a health questionnaire. Participants will also complete a food frequency questionnaire to assess food/drink intake over the past week. Height will be assessed via a calibrated stadiometer and weight will be assessed by calibrated digital scale in street clothes and without shoes. Participants will be reminded to abstain from consuming high calorie foods/drinks through the end of the day of the 24-hr follow-up session.

After the baseline session, participants will be randomized to either a high calorie food retrieval + high calorie food extinction (R-E training) group or to a non-food retrieval + high calorie food extinction (extinction control) group at the next two sessions.

R-E/EXTINCTION TRAINING SESSIONS: Participants will return to the lab on the next two consecutive days after the baseline session to engage in food-related retrieval + 60-min extinction training for high calorie foods (R-E training group) or non-food-related retrieval + 60-min extinction training for high calorie foods (extinction control group). These two sessions will last approximately 2.5-hr each and will be identical in their procedures. Similar to the baseline session, participants will first be interviewed to report past 24-hr food/drink intake and past 24-hr health-related behaviors including nicotine, alcohol, caffeine, cannabis, and other substance use, medication use, sleep, and physical activity. After the 10-min acclimation period, participants will complete baseline assessments of hunger and craving (self-report, heart rate, skin conductance, salivation). During the R-E and extinction control training, participants will first observe retrieval cues: either the same sequence of high calorie food cues observed at the baseline session (R-E training group) or a sequence of non-food-related cues (extinction control group). After 10-min of rest following retrieval, all participants will engage in 60-min of high calorie food extinction training (see complete details in the "TASK DESCRIPTION" section below). Measures of heart rate, skin conductance, and salivation will be collected throughout extinction training. Finally, participants will repeat assessments of negative and positive affect and will be weighed.

FOLLOW-UP SESSIONS: Follow-up sessions will occur 24-hr, 2-week, and 1- and 3-month after the second R-E/extinction training session and will last approximately two hr each. Sessions will begin with an interview to assess recent food and drink intake and past 24-hr health behaviors. After 10-min of acclimation, participants will complete baseline craving, hunger, and psychophysiological (heart rate, skin conductance, salivation) measures, a food cue-reactivity task, and weight measurement. Similar to prior sessions, heart rate, skin conductance, and salivation will be collected throughout the food cue-reactivity task. Participants will also repeat assessments of motivation to lose weight, state food craving, dietary restraint and disinhibited eating, impulsivity, negative and positive affect, physical activity, eating behavior, and reward-based eating drive at follow-up sessions. Participants will complete a past-week food frequency questionnaire at the 2-week, 1-month, and 3-month follow-up sessions as well as the bogus taste test at 1- and 3-month follow-up (identical to the baseline session). Participants will be weighed at the end of every session.

EMA: Half of the participants involved in this clinical trial (n=75; starting in Year 3 of the funding period) will engage in EMA to collect data on naturally-occurring food cues, eating context (e.g., presence of others, eating context), food craving, hunger, negative and positive affect, and food intake via EMA. Data will be collected through a web-based app developed through the Office of Academic Computing at the University of Pittsburgh. Data collection will occur in three measurement bursts over three consecutive days (a) ~4-6 days before baseline, and between (b) 24-hr and 2-week, and (c) 2-week and 1-month follow-up. Participants will be asked to respond to (a) 'random,' (b) 'time-contingent,' and (c) 'event-contingent' prompts. Random assessments will occur at random times over the 3-day measurement bursts and time-contingent assessments will occur at fixed times each day, including beginning and end of day prompts sent at participant-preferred times. On average, participants will be prompted five times daily on each of the three EMA days. Participants will be instructed to initiate event-contingent assessments when a predefined event occurs, including eating or craving food. To encourage compliance, participants will be compensated per EMA entry and a daily bonus when all prompted entries are completed.

TASK DESCRIPTION

FOOD CUE-REACTIVITY TASK: The food cue-reactivity task is a computerized task programmed using E-Prime software. At the baseline session, participants will observe 30 high calorie pictorial food cues on the computer in a 5-min cue sequence. At each follow-up session participants will observe the same 5-min high calorie food cue sequence observed at the baseline session plus an additional novel 5-min high calorie food cue sequence to assess the generalizability of R-E/extinction control training to novel food cues. During a 5-min cue sequence, participants will observe a pictorial food cue on the computer screen for 8-s each, with a 2-s delay between pictorial cues, resulting in 5-min of high calorie pictorial food cue presentation at baseline and 10-min at each follow-up session. Self-report craving will be assessed after the first 2-min of cue presentation and again at the end of the cue sequence. The first self-report craving assessment will occur at 2-min into the cue sequence to coincide with the salivation measure that will occur across the same 2-min (the Strongin-Hinsie Peck procedure). Heart rate and skin conductance will be assessed continuously throughout 5-min cue sequences.

R-E/EXTINCTION TRAINING CONTROL: On both training days, participants will observe retrieval cues: either the same 5-min sequence of high calorie pictorial food cues observed during the food cue-reactivity task at the baseline session (R-E training group) or 5-min of non-food-related cues (extinction control group). After 10-min of rest following retrieval, all participants will engage in 60-min of high calorie food extinction training. Extinction training will involve 12, 5-min high calorie food cue sequences: 6 pictorial and 6 real food cue sequences. Pictorial food cue sequences will involve timing that is identical to pictorial food cue sequences at the other sessions: participants will observe a pictorial food cue on the computer screen for 8-s each, with a 2-s delay between pictorial cues. Real food cues will be individualized for each participant, reflecting foods with the highest palatability ratings provided during phone screening. During 5-min real food cue sequences, participants will be instructed to remove the food from its bowl and to observe, handle, smell, bring the food to their lips, and imagine eating the food. Self-reported craving will be assessed at the same time points as during the 5-min cue sequences of food cue-reactivity tasks at other sessions: 2-min into cue sequences and again at the end of 5-min cue sequences. Salivation will not be assessed during the 60-min of extinction training to reduce participant burden and ensure that extinction training has its intended effects (i.e., to avoid interference of collecting numerous saliva measures on the effectiveness of extinction training). Heart rate and skin conductance will be measured continuously throughout the 60-min of extinction training.

BOGUS TASTE TEST: The validated bogus taste test will be used to assess in-lab food intake at the baseline session and the 1- and 3-month follow-up sessions. During the bogus taste test, participants will be provided four, 12-ounce bowls filled with the four high calorie foods with the highest palatability ratings provided during phone screening. Participants will be instructed to take at least one bite of each food and answer taste perception questions about those foods. Participants will be instructed that they have 10-min to complete this task and can eat leftover foods in any remaining time. Unknown to participants, food bowls will be weighed pre- and post-task to assess the amount of food consumed. Food consumed (g) will be converted into energy intake (calories) for analysis.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 18-59 years
* Body mass index ≥25.0, indicating overweight/obesity
* Interested in losing weight
* Adequate liking of ≥4 foods to be presented during extinction training
* Willing to complete the following necessary study procedures: (1) eat study foods during taste test, (2) have heart rate sensors placed on skin, (3) abstain from alcohol, cannabis, benzodiazepines, opiates, or other illegal substances starting at midnight before each session, (4) attend sessions at the same time each day and starting with Session 1 on a Monday or Tuesday, and (5) abstain from consuming high calorie foods/drinks across the first 4 sessions

EXCLUSION CRITERIA:

* Engaged in a weight loss treatment/program or involved in another research study providing treatment/intervention for weight loss
* Participation in a food cue-reactivity pilot study that used procedures similar to those of the current study (e.g., food cue-reactivity task, bogus taste test)
* Diabetes diagnosis
* Initiation of thyroid-related medications or, for women, initiation of new birth control medication, an implant, or intrauterine device in the past 3 months
* Regular use of benzodiazepines (i.e., >5 times in the past 30 days)
* Use of weight- or appetite-affecting medication
* Currently receiving treatment for an eating disorder
* Bariatric surgery in the past 3 years
* Food allergies or restrictions over the next 4 months preventing consumption of foods presented during lab tasks
* Has a pacemaker implant
* For women: currently pregnant or planning to become pregnant in the next 4 months
* For women: currently breastfeeding with >50% of baby's/child's nutrition coming from breast milk

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Self-Report State Food Craving Response to High Calorie Food Cues at 24-hr Follow-up | current; assess change from baseline vs. 24-hr follow-up
  Self-reported state food craving in response to high calorie foods presented during the study will be assessed using the 3-item Intense Desire to Eat subscale of the Food Cravings Questionnaire-State (with modified numerical anchors to increase variability in responding). Participants will report the craving they are experiencing "right now, at this very moment" on a 0 (strongly disagree) to 100 (strongly agree) Likert rating scale. Mean scores will be calculated by averaging across ratings for a possible range of scores between 0 and 100, with higher scores reflecting greater self-reported craving.
Mean Change from Baseline in Self-Report State Food Craving Response to High Calorie Food Cues at 2-week Follow-up | current; assess change from baseline vs. 2-week follow-up
  Self-reported state food craving in response to high calorie foods presented during the study will be assessed using the 3-item Intense Desire to Eat subscale of the Food Cravings Questionnaire-State (with modified numerical anchors to increase variability in responding). Participants will report the craving they are experiencing "right now, at this very moment" on a 0 (strongly disagree) to 100 (strongly agree) Likert rating scale. Mean scores will be calculated by averaging across ratings for a possible range of scores between 0 and 100, with higher scores reflecting greater self-reported craving.
Mean Change from Baseline in Self-Report State Food Craving Response to High Calorie Food Cues at 1-month Follow-up | current; assess change from baseline vs. 1-month follow-up
  Self-reported state food craving in response to high calorie foods presented during the study will be assessed using the 3-item Intense Desire to Eat subscale of the Food Cravings Questionnaire-State (with modified numerical anchors to increase variability in responding). Participants will report the craving they are experiencing "right now, at this very moment" on a 0 (strongly disagree) to 100 (strongly agree) Likert rating scale. Mean scores will be calculated by averaging across ratings for a possible range of scores between 0 and 100, with higher scores reflecting greater self-reported craving.
Mean Change from Baseline in Self-Report State Food Craving Response to High Calorie Food Cues at 3-month Follow-up | current; assess change from baseline vs. 3-month follow-up
  Self-reported state food craving in response to high calorie foods presented during the study will be assessed using the 3-item Intense Desire to Eat subscale of the Food Cravings Questionnaire-State (with modified numerical anchors to increase variability in responding). Participants will report the craving they are experiencing "right now, at this very moment" on a 0 (strongly disagree) to 100 (strongly agree) Likert rating scale. Mean scores will be calculated by averaging across ratings for a possible range of scores between 0 and 100, with higher scores reflecting greater self-reported craving.
Differences between R-E Training Group and Extinction Control Group in Self-Report State Food Craving Response to High Calorie Food Cues at 24-hr Follow-up | current; assess differences between groups at 24-hr follow-up
  Self-reported state food craving in response to high calorie foods presented during the study will be assessed using the 3-item Intense Desire to Eat subscale of the Food Cravings Questionnaire-State (with modified numerical anchors to increase variability in responding). Participants will report the craving they are experiencing "right now, at this very moment" on a 0 (strongly disagree) to 100 (strongly agree) Likert rating scale. Mean scores will be calculated by averaging across ratings for a possible range of scores between 0 and 100, with higher scores reflecting greater self-reported craving.
Differences between R-E Training Group and Extinction Control Group in Self-Report State Food Craving Response to High Calorie Food Cues at 2-week Follow-up | current; assess differences between groups at 2-week follow-up
  Self-reported state food craving in response to high calorie foods presented during the study will be assessed using the 3-item Intense Desire to Eat subscale of the Food Cravings Questionnaire-State (with modified numerical anchors to increase variability in responding). Participants will report the craving they are experiencing "right now, at this very moment" on a 0 (strongly disagree) to 100 (strongly agree) Likert rating scale. Mean scores will be calculated by averaging across ratings for a possible range of scores between 0 and 100, with higher scores reflecting greater self-reported craving.
Differences between R-E Training Group and Extinction Control Group in Self-Report State Food Craving Response to High Calorie Food Cues at 1-month Follow-up | current; assess differences between groups at 1-month follow-up
  Self-reported state food craving in response to high calorie foods presented during the study will be assessed using the 3-item Intense Desire to Eat subscale of the Food Cravings Questionnaire-State (with modified numerical anchors to increase variability in responding). Participants will report the craving they are experiencing "right now, at this very moment" on a 0 (strongly disagree) to 100 (strongly agree) Likert rating scale. Mean scores will be calculated by averaging across ratings for a possible range of scores between 0 and 100, with higher scores reflecting greater self-reported craving.
Differences between R-E Training Group and Extinction Control Group in Self-Report State Food Craving Response to High Calorie Food Cues at 3-month Follow-up | current; assess differences between groups at 3-month follow-up
  Self-reported state food craving in response to high calorie foods presented during the study will be assessed using the 3-item Intense Desire to Eat subscale of the Food Cravings Questionnaire-State (with modified numerical anchors to increase variability in responding). Participants will report the craving they are experiencing "right now, at this very moment" on a 0 (strongly disagree) to 100 (strongly agree) Likert rating scale. Mean scores will be calculated by averaging across ratings for a possible range of scores between 0 and 100, with higher scores reflecting greater self-reported craving.
Mean Change from Baseline in Heart Rate Response to High Calorie Food Cues at 24-hr Follow-up | current; assess change from baseline vs. 24-hr follow-up
  Heart rate data will be collected using electrodes affixed below the ribcage and clavicle. MindWare Technologies hardware will collect continuous heart rate data during the presentation of high calorie food cues. Heart rate will be measured on a continuous scale with higher heart rate reflecting greater reactivity to high calorie food cues.
Mean Change from Baseline in Heart Rate Response to High Calorie Food Cues at 2-week Follow-up | current; assess change from baseline vs. 2-week follow-up
  Heart rate data will be collected using electrodes affixed below the ribcage and clavicle. MindWare Technologies hardware will collect continuous heart rate data during the presentation of high calorie food cues. Heart rate will be measured on a continuous scale with higher heart rate reflecting greater reactivity to high calorie food cues.
Mean Change from Baseline in Heart Rate Response to High Calorie Food Cues at 1-month Follow-up | current; assess change from baseline vs. 1-month follow-up
  Heart rate data will be collected using electrodes affixed below the ribcage and clavicle. MindWare Technologies hardware will collect continuous heart rate data during the presentation of high calorie food cues. Heart rate will be measured on a continuous scale with higher heart rate reflecting greater reactivity to high calorie food cues.
Mean Change from Baseline in Heart Rate Response to High Calorie Food Cues at 3-month Follow-up | current; assess change from baseline vs. 3-month follow-up
  Heart rate data will be collected using electrodes affixed below the ribcage and clavicle. MindWare Technologies hardware will collect continuous heart rate data during the presentation of high calorie food cues. Heart rate will be measured on a continuous scale with higher heart rate reflecting greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Heart Rate Response to High Calorie Food Cues at 24-hr Follow-up | current; assess differences between groups at 24-hr follow-up
  Heart rate data will be collected using electrodes affixed below the ribcage and clavicle. MindWare Technologies hardware will collect continuous heart rate data during the presentation of high calorie food cues. Heart rate will be measured on a continuous scale with higher heart rate reflecting greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Heart Rate Response to High Calorie Food Cues at 2-week Follow-up | current; assess differences between groups at 2-week follow-up
  Heart rate data will be collected using electrodes affixed below the ribcage and clavicle. MindWare Technologies hardware will collect continuous heart rate data during the presentation of high calorie food cues. Heart rate will be measured on a continuous scale with higher heart rate reflecting greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Heart Rate Response to High Calorie Food Cues at 1-month Follow-up | current; assess differences between groups at 1-month follow-up
  Heart rate data will be collected using electrodes affixed below the ribcage and clavicle. MindWare Technologies hardware will collect continuous heart rate data during the presentation of high calorie food cues. Heart rate will be measured on a continuous scale with higher heart rate reflecting greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Heart Rate Response to High Calorie Food Cues at 3-month Follow-up | current; assess differences between groups at 3-month follow-up
  Heart rate data will be collected using electrodes affixed below the ribcage and clavicle. MindWare Technologies hardware will collect continuous heart rate data during the presentation of high calorie food cues. Heart rate will be measured on a continuous scale with higher heart rate reflecting greater reactivity to high calorie food cues.
Mean Change from Baseline in Skin Conductance Response to High Calorie Food Cues at 24-hr Follow-up | current; assess change from baseline vs. 24-hr follow-up
  Skin conductance data will be collected using two electrodes placed on the palm of the hand. MindWare Technologies hardware will collect continuous skin conductance data during the presentation of high calorie food cues with greater skin conductance reflecting greater reactivity to high calorie food cues.
Mean Change from Baseline in Skin Conductance Response to High Calorie Food Cues at 2-week Follow-up | current; assess change from baseline vs. 2-week follow-up
  Skin conductance data will be collected using two electrodes placed on the palm of the hand. MindWare Technologies hardware will collect continuous skin conductance data during the presentation of high calorie food cues with greater skin conductance reflecting greater reactivity to high calorie food cues.
Mean Change from Baseline in Skin Conductance Response to High Calorie Food Cues at 1-month Follow-up | current; assess change from baseline vs. 1-month follow-up
  Skin conductance data will be collected using two electrodes placed on the palm of the hand. MindWare Technologies hardware will collect continuous skin conductance data during the presentation of high calorie food cues with greater skin conductance reflecting greater reactivity to high calorie food cues.
Mean Change from Baseline in Skin Conductance Response to High Calorie Food Cues at 3-month Follow-up | current; assess change from baseline vs. 3-month follow-up
  Skin conductance data will be collected using two electrodes placed on the palm of the hand. MindWare Technologies hardware will collect continuous skin conductance data during the presentation of high calorie food cues with greater skin conductance reflecting greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Skin Conductance Response to High Calorie Food Cues at 24-hr Follow-up | current; assess differences between groups at 24-hr follow-up
  Skin conductance data will be collected using two electrodes placed on the palm of the hand. MindWare Technologies hardware will collect continuous skin conductance data during the presentation of high calorie food cues with greater skin conductance reflecting greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Skin Conductance Response to High Calorie Food Cues at 2-week Follow-up | current; assess differences between groups at 2-week follow-up
  Skin conductance data will be collected using two electrodes placed on the palm of the hand. MindWare Technologies hardware will collect continuous skin conductance data during the presentation of high calorie food cues with greater skin conductance reflecting greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Skin Conductance Response to High Calorie Food Cues at 1-month Follow-up | current; assess differences between groups at 1-month follow-up
  Skin conductance data will be collected using two electrodes placed on the palm of the hand. MindWare Technologies hardware will collect continuous skin conductance data during the presentation of high calorie food cues with greater skin conductance reflecting greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Skin Conductance Response to High Calorie Food Cues at 3-month Follow-up | current; assess differences between groups at 3-month follow-up
  Skin conductance data will be collected using two electrodes placed on the palm of the hand. MindWare Technologies hardware will collect continuous skin conductance data during the presentation of high calorie food cues with greater skin conductance reflecting greater reactivity to high calorie food cues.
Mean Change from Baseline in Salivation Response to High Calorie Food Cues at 24-hr Follow-up | current; assess change from baseline vs. 24-hr follow-up
  Salivation in response to observing high calorie food cues will be collected using three cotton dental rolls (two placed buccally and one placed beneath the tongue) for 2-min segments according to the Strongin-Hinsie Peck method. The dental rolls will be weighed (in grams) to assess the amount of saliva produced. Greater salivation (indicated by heavier weight of dental rolls) will indicate greater reactivity to high calorie food cues.
Mean Change from Baseline in Salivation Response to High Calorie Food Cues at 2-week Follow-up | current; assess change from baseline vs. 2-week follow-up
  Salivation in response to observing high calorie food cues will be collected using three cotton dental rolls (two placed buccally and one placed beneath the tongue) for 2-min segments according to the Strongin-Hinsie Peck method. The dental rolls will be weighed (in grams) to assess the amount of saliva produced. Greater salivation (indicated by heavier weight of dental rolls) will indicate greater reactivity to high calorie food cues.
Mean Change from Baseline in Salivation Response to High Calorie Food Cues at 1-month Follow-up | current; assess change from baseline vs. 1-month follow-up
  Salivation in response to observing high calorie food cues will be collected using three cotton dental rolls (two placed buccally and one placed beneath the tongue) for 2-min segments according to the Strongin-Hinsie Peck method. The dental rolls will be weighed (in grams) to assess the amount of saliva produced. Greater salivation (indicated by heavier weight of dental rolls) will indicate greater reactivity to high calorie food cues.
Mean Change from Baseline in Salivation Response to High Calorie Food Cues at 3-month Follow-up | current; assess change from baseline vs. 3-month follow-up
  Salivation in response to observing high calorie food cues will be collected using three cotton dental rolls (two placed buccally and one placed beneath the tongue) for 2-min segments according to the Strongin-Hinsie Peck method. The dental rolls will be weighed (in grams) to assess the amount of saliva produced. Greater salivation (indicated by heavier weight of dental rolls) will indicate greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Salivation Response to High Calorie Food Cues at 24-hr Follow-up | current; assess differences between groups at 24-hr follow-up
  Salivation in response to observing high calorie food cues will be collected using three cotton dental rolls (two placed buccally and one placed beneath the tongue) for 2-min segments according to the Strongin-Hinsie Peck method. The dental rolls will be weighed (in grams) to assess the amount of saliva produced. Greater salivation (indicated by heavier weight of dental rolls) will indicate greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Salivation Response to High Calorie Food Cues at 2-week Follow-up | current; assess differences between groups at 2-week follow-up
  Salivation in response to observing high calorie food cues will be collected using three cotton dental rolls (two placed buccally and one placed beneath the tongue) for 2-min segments according to the Strongin-Hinsie Peck method. The dental rolls will be weighed (in grams) to assess the amount of saliva produced. Greater salivation (indicated by heavier weight of dental rolls) will indicate greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Salivation Response to High Calorie Food Cues at 1-month Follow-up | current; assess differences between groups at 1-month follow-up
  Salivation in response to observing high calorie food cues will be collected using three cotton dental rolls (two placed buccally and one placed beneath the tongue) for 2-min segments according to the Strongin-Hinsie Peck method. The dental rolls will be weighed (in grams) to assess the amount of saliva produced. Greater salivation (indicated by heavier weight of dental rolls) will indicate greater reactivity to high calorie food cues.
Differences between R-E Training Group and Extinction Control Group in Salivation Response to High Calorie Food Cues at 3-month Follow-up | current; assess differences between groups at 3-month follow-up
  Salivation in response to observing high calorie food cues will be collected using three cotton dental rolls (two placed buccally and one placed beneath the tongue) for 2-min segments according to the Strongin-Hinsie Peck method. The dental rolls will be weighed (in grams) to assess the amount of saliva produced. Greater salivation (indicated by heavier weight of dental rolls) will indicate greater reactivity to high calorie food cues.

SECONDARY OUTCOMES:
Mean Change from Baseline in Consumption of High Calorie Foods/Drinks at 2-week Follow-up | current; assess change from baseline vs. 2-week follow-up
  Food/drink intake will be assessed using a self-report food frequency questionnaire: the Diet History Questionnaire (DHQ) III. The DHQ III will be modified to: (a) assess high calorie foods and drinks targeted by the intervention, and (b) assess food/drink intake over the past week. Higher scores on the DHQ III will indicate greater intake of high calorie foods/drinks.
Mean Change from Baseline in Consumption of High Calorie Foods/Drinks at 1-month Follow-up | current; assess change from baseline vs. 1-month follow-up
  Food/drink intake will be assessed using a self-report food frequency questionnaire: the Diet History Questionnaire (DHQ) III. The DHQ III will be modified to: (a) assess high calorie foods and drinks targeted by the intervention, and (b) assess food/drink intake over the past week. Higher scores on the DHQ III will indicate greater intake of high calorie foods/drinks.
Mean Change from Baseline in Consumption of High Calorie Foods/Drinks at 3-month Follow-up | current; assess change from baseline vs. 3-month follow-up
  Food/drink intake will be assessed using a self-report food frequency questionnaire: the Diet History Questionnaire (DHQ) III. The DHQ III will be modified to: (a) assess high calorie foods and drinks targeted by the intervention, and (b) assess food/drink intake over the past week. Higher scores on the DHQ III will indicate greater intake of high calorie foods/drinks.
Differences between R-E Training Group and Extinction Control Group in Consumption of High Calorie Foods/Drinks at 2-week Follow-up | current; assess differences between groups at 2-week follow-up
  Food/drink intake will be assessed using a self-report food frequency questionnaire: the Diet History Questionnaire (DHQ) III. The DHQ III will be modified to: (a) assess high calorie foods and drinks targeted by the intervention, and (b) assess food/drink intake over the past week. Higher scores on the DHQ III will indicate greater intake of high calorie foods/drinks.
Differences between R-E Training Group and Extinction Control Group in Consumption of High Calorie Foods/Drinks at 1-month Follow-up | current; assess differences between groups at 1-month follow-up
  Food/drink intake will be assessed using a self-report food frequency questionnaire: the Diet History Questionnaire (DHQ) III. The DHQ III will be modified to: (a) assess high calorie foods and drinks targeted by the intervention, and (b) assess food/drink intake over the past week. Higher scores on the DHQ III will indicate greater intake of high calorie foods/drinks.
Differences between R-E Training Group and Extinction Control Group in Consumption of High Calorie Foods/Drinks at 3-month Follow-up | current; assess differences between groups at 3-month follow-up
  Food/drink intake will be assessed using a self-report food frequency questionnaire: the Diet History Questionnaire (DHQ) III. The DHQ III will be modified to: (a) assess high calorie foods and drinks targeted by the intervention, and (b) assess food/drink intake over the past week. Higher scores on the DHQ III will indicate greater intake of high calorie foods/drinks.
Mean Change from Baseline in Body Weight at 2-week Follow-up | current; assess change from baseline vs. 2-week follow-up
  Participants will be weighed while in street clothes and without shoes using a calibrated digital scale.
Mean Change from Baseline in Body Weight at 1-month Follow-up | current; assess change from baseline vs. 1-month follow-up
  Participants will be weighed while in street clothes and without shoes using a calibrated digital scale.
Mean Change from Baseline in Body Weight at 3-month Follow-up | current; assess change from baseline vs. 3-month follow-up
  Participants will be weighed while in street clothes and without shoes using a calibrated digital scale.
Differences between R-E Training Group and Extinction Control Group in Body Weight at 2-week Follow-up | current; assess differences between groups at 2-week follow-up
  Participants will be weighed while in street clothes and without shoes using a calibrated digital scale.
Differences between R-E Training Group and Extinction Control Group in Body Weight at 1-month Follow-up | current; assess differences between groups at 1-month follow-up
  Participants will be weighed while in street clothes and without shoes using a calibrated digital scale.
Differences between R-E Training Group and Extinction Control Group in Body Weight at 3-month Follow-up | current; assess differences between groups at 3-month follow-up
  Participants will be weighed while in street clothes and without shoes using a calibrated digital scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Germeroth, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures, along with data dictionaries, will be made available without cost to researchers and analysts in the general scientific community. Data will be provided in statistical formats including Statistical Package for Social Sciences (SPSS) file format and will represent the final research data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available no later than the acceptance for publication of the main findings from the final data set. Data will be available indefinitely through a data archive.
Access Criteria: Any researcher or analyst in the scientific community will have access to the data via a database and management website such as Mendeley Data.